CLINICAL TRIAL: NCT07309822
Title: Observational Prospective Study to Assess the Safety and Effectiveness of Beltaven® in Patients With Allergy to Apis Mellifera, Polistes Dominula or Vespula Spp
Brief Title: Study to Assess the Safety and Effectiveness of Beltaven® in Patients With Allergy to Apis Mellifera, Polistes Dominula or Vespula Spp.
Status: Recruiting | Type: Observational
Sponsor: Probelte Pharma S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-VEN-2023-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-interventional Study to Assess the Safety and Effectiveness Profile of a SCIT Therapy With Beltaven® With Apis mellifera, Polistes dominula or Vespula spp. allergic patients

DETAILED DESCRIPTION:
This prospective open multi-centre non-interventional study assess the safety and effectiveness profile of the subcutaneous allergen-specific immunotherapy with Beltaven in Apis mellifera, Polistes dominula or Vespula spp (children and adults) in routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 years or older at the time of study inclusion.
* Written informed consent, duly signed and dated by the patient or by the legal representative in the case of minors.
* Assent form duly signed and dated by the minor, when applicable.
* Patients with allergy to Apis mellifera, Vespula spp., or Polistes dominula who have experienced a systemic reaction following a hymenoptera sting, either with involvement of multiple organs or exclusively cutaneous.
* Positive intradermal test (mean wheal diameter ≥ 5 mm) with Beltaven® diagnostic (allergenic extract of Apis mellifera, Vespula spp., or Polistes dominula).
* Positive specific IgE test from class 1 onwards (≥ 0.35 kUA/L).
* Patients willing to receive immunotherapy with Beltaven®.

Exclusion Criteria:

* Patients with severe cardiovascular diseases, active malignant neoplasms or malignancies in remission within the last 5 years, non-stabilized systemic or organ-specific autoimmune diseases, severe mental disorders, or other relevant chronic diseases that may interfere with the study results.
* Patients with known allergy to any of the vaccine excipients.
* Pregnant patients, patients planning to become pregnant during the study period, or breastfeeding patients.
* Patients who have received hymenoptera immunotherapy within the 5 years prior to inclusion or during the study.
* Patients who are to receive immunotherapy with another specific allergen different from the investigational treatment during the study period.
* Patients with confirmed sensitization to two or more hymenoptera species as demonstrated by CAP inhibition testing.
* Patients with thrombocytopenic purpura and vasculitis, rhabdomyolysis, or renal failure.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 14 years with allergy to hymenoptera venom (Apis mellifera, Vespula spp., or Polistes dominula)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical effectiveness of Beltaven® administered subcutaneously following a 3-week cluster dosing regimen | 9 months
  Proportion of patients who show tolerance (absence of systemic reaction) to the controlled sting challenge test conducted during the challenge visit, or to an accidental sting in a rural setting during the continuation treatment period

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - Hospital Universitario Vall d' Hebron, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Xarxa Assistencial I Universitària de Manresa, Barcelona
  - Hospital General Universitario de Castellón, Castellon
  - Hospital General la Mancha Centro, Ciudad Real
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Santa Caterina de Girona, Girona
  - Hospital Universitario Santa María de Lleida, Lleida
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Vega Baja, Orihuela